CLINICAL TRIAL: NCT02342925
Title: A Study of the Effect of RG1662 on Metformin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: WP29394; 2014-001851-21 (EudraCT Number)
Record Dates: First submitted 2015-01-07; First posted 2015-01-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Iohexol; Metformin

ARMS (2):
- RG1662 plus metformin (Experimental)
  Interventions: Other: Omnipaque 300; Drug: RG1662; Drug: metformin
- metformin alone (Experimental)
  Interventions: Other: Omnipaque 300; Drug: metformin

INTERVENTIONS:
Other: Omnipaque 300 — 647 mg/mL of iohexol, equivalent to 300 mg/mL of iodine, used for assessment of glomerular function and other measure of renal function
Drug: RG1662 — Oral administration twice daily
  Arms: RG1662 plus metformin
Drug: metformin — Single 850 mg dose of metformin

SUMMARY:
This single-center, non-randomized, open-label, two treatment, two period, fixed sequence crossover study will investigate the effect of RG1662 treatment on the activity of key renal transporters in healthy male and female participants using metformin. The effect of RG1662 on other renal function parameters will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants, aged 18 to 60 years, inclusive
* A body mass index between 18 to 32 kg/m2, inclusive
* Informed consent and agreement to comply with study restrictions

Exclusion Criteria:

* A history of epilepsy, convulsions or significant head injury
* Significant history of drug allergy or a known hypersensitivity to any of the ingredients of any of the study treatments
* Pregnant or lactating
* Impaired renal function or clinically relevant hematuria
* A history of lactic acidosis, or risk factors for lactic acidosis
* Any other clinically relevant abnormalities, concomitant diseases or ongoing medical conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of metformin derived from plasma and urine concentrations of metformin: area under the concentration-time curve (AUC), maximum concentration (Cmax), renal clearance (CLr) [composite outcome measure] | Up to 9 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters derived from plasma concentrations of RG1662: AUC, Cmax, time to maximum concentration (Tmax), and minimum concentration (Ctrough)[composite outcome measure] | Up to 9 weeks
Pharmacodynamics: renal function measured by derivation of glomerular filtration rate (GFR) from plasma concentrations of iohexol. | Up to 9 weeks
Incidence of adverse events (AEs) | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leeds, United Kingdom